CLINICAL TRIAL: NCT03879824
Title: Radial Versus Femoral Secondary Access in Patients Undergoing Transcatheter Aortic Valve Implantation (R-TAVI): A Randomized Pilot Study
Brief Title: Radial Versus Femoral Secondary Access During TAVI
Acronym: R-TAVI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI and co-investigators would like to terminate the study given challenges with patient enrollment.
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Rahul Sharma, Assistant Director Structural Heart & Valve Center/Assistant Professor of Medicine Virginia Tech Carilion School of Medicine, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2611
Record Dates: First submitted 2018-12-11; First posted 2019-03-19 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Aortic Stenosis; Aortic Valve Disease; Vascular Access Complication
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial Artery Secondary Access During TAVI (Experimental): Patients randomized to this arm will undergo primary access for valve placement through the femoral artery and will have secondary vascular access for placement of the pigtail catheter through the radial artery (right radial artery only) during their transcatheter aortic valve implantation (TAVI)
  The active intervention in this arm of the study is secondary radial artery access during TAVI
  Interventions: Procedure: Secondary Radial Artery Access
- Femoral Artery Secondary Access During TAVI (Active Comparator): Patients randomized to this arm will undergo primary access for valve placement through the femoral artery and will have secondary vascular access for placement of the pigtail catheter through the contralateral femoral artery artery during their transcatheter aortic valve implantation (TAVI)
  The active intervention in this arm of the study is secondary femoral artery access during TAVI
  Interventions: Procedure: Secondary Femoral Artery Access

INTERVENTIONS:
Procedure: Secondary Radial Artery Access — Patients undergoing transcatheter aortic valve implantation (TAVI) will receive secondary arterial access via percutaneous access of the right radial artery for the purpose of insertion of a standard pigtail catheter for aortic route angiography during TAVI.
  Arms: Radial Artery Secondary Access During TAVI
Procedure: Secondary Femoral Artery Access — Patients undergoing transcatheter aortic valve implantation (TAVI) will receive secondary arterial access via percutaneous access of the contralateral femoral artery for the purpose of insertion of a standard pigtail catheter for aortic route angiography during TAVI.
  Arms: Femoral Artery Secondary Access During TAVI

SUMMARY:
The R-TAVI study is a randomized pilot study examining the use of the right radial artery versus the femoral artery for secondary vascular access during transcatheter aortic valve implantation (TAVI).

DETAILED DESCRIPTION:
The R-TAVI study is a prospective, single institution, pilot study in which eligible TAVI patients will be randomized pre-procedurally to receive either secondary radial artery (RA) access or femoral artery (FA) access during TAVI. Our study will take place over a projected 18 month enrollment period.

ELIGIBILITY:
Inclusion Criteria:

1) Patient meets eligibility for TAVR as decided upon by pre-TAVR testing (Echo, cardiac catheterization, CTA TAVR, 2 CT surgical consults, heart team discussion). 2) Undergoing TAVR procedure and follow-up at Carilion Clinic Cardiology Roanoke Memorial Hospital (CRMH) 3) Patient's secondary vascular access can be performed femorally OR radially, as determined by TAVR operator after review of pre-TAVR CT scan imaging.

4) Interventional Cardiologist performing the TAVR agrees to consider patient for enrollment.

5) Patient provides consent 6) Age ≥ 18 years old 7) No evidence of precluding arterial disease of both femoral arteries 8) No evidence of precluding arterial disease of right radial and subclavian arteries 9) Must have palpable pulses in both radial arteries

Exclusion Criteria:

1. Review of pre-TAVR CT scan imaging deems patient unsuitable for radial OR femoral secondary access based on presence of excessive calcification, stenosis, or tortuosity of the femoral, subclavian, or innominate arteries.
2. Valve implantation (primary access) planned via alternative vascular access (trans-caval, axillary, carotid, direct aortic, trans-apical)-as determined by implanting Interventional Cardiologist/TAVR operator.
3. Prior coronary artery bypass graft surgery in which a radial artery graft was harvested and used as a conduit.
4. Patients on hemodialysis OR with arteriovenous fistulas.
5. Interventional Cardiologist performing the TAVR declines patient consideration in the study.
6. Patient declines consent.
7. Urgent or emergent TAVI cases
8. Patient is already participating in another clinical research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Number of Patients who Develop Death, MI, Stroke, and ACUITY major bleeding from the start of the TAVI procedure until hospital discharge | At time of hospital discharge (ranges from 24 hours post procedure - 72 hours post procedure)
  We will report the number of patients who develop death, myocardial infarction, stroke, and/or ACUITY major bleeding definitions from the start of the TAVI procedure to the the time of patient's hospital discharge after undergoing the TAVI procedure.
  The time of hospital discharge ranges from 24 -72 hours after TAVI procedure, depending on the patient's course of recovery.
  This will be reported as a composite incidence of death, MI, stroke and ACUITY major bleeding.
Number of Patients who Develop Death, MI, Stroke, and ACUITY major bleeding within 30 days post TAVI procedure | Procedure start to 30-day follow-up.
  We will report the number of patients who develop death, myocardial infarction, stroke, and/or ACUITY major bleeding definitions from the start of the TAVI procedure to the the time of their 30-day post TAVI follow up
  This will be reported as a 30-day composite incidence of death, MI, stroke and ACUITY major bleeding.

SECONDARY OUTCOMES:
Number of patients who successfully undergo completion ileofemoral angiography of the valve implantation access site via the randomized secondary arterial access site | Intra-procedural metric
Number of patients who underwent successful endovascular intervention to the valve implantation ileofemoral access site via the randomized secondary access point | Intra-procedural metric
Radiation Dose (in minutes of fluoroscopy time) | Intra-procedural metric
Radiation Dose (in milligrays, mGy) | Intra-procedural metric
Procedure Start-Stop Time (minutes) | Intra-procedural metric
Number of patients requiring conversion to secondary femoral access from secondary radial access | Intra-procedural metric
Number of patients who developed a major vascular complications, as defined by the 2nd Valve Academic Research Consortium (VARC-2) Criteria from the start of the TAVI procedure until hospital discharge | At time of hospital discharge (ranges from 24 hours post procedure - 72 hours post procedure)
  The time of hospital discharge ranges from 24 -72 hours after TAVI procedure, depending on the patient's course of recovery.
Number of patients who developed a major vascular complications, as defined by the 2nd Valve Academic Research Consortium (VARC-2) Criteria within 30 days post TAVI procedure | At 30 Day Follow-Up
Number of patients who developed a minor vascular complications, as defined by the 2nd Valve Academic Research Consortium (VARC-2) Criteria from the start of the TAVI procedure until hospital discharge | At time of hospital discharge (ranges from 24 hours post procedure - 72 hours post procedure)
  The time of hospital discharge ranges from 24 -72 hours after TAVI procedure, depending on the patient's course of recovery.
Number of patients who developed a minor vascular complications, as defined by the 2nd Valve Academic Research Consortium (VARC-2) Criteria within 30 days post TAVI procedure | At 30 Day Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Sharma, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No